CLINICAL TRIAL: NCT04179110
Title: A Phase II Trial of Pembrolizumab and Ramucirumab in Patients With Progressive Transitional Cell Carcinoma After Treatment With an Immune Checkpoint Inhibitor
Brief Title: Study of Pembrolizumab and Ramucirumab in Pts With Progressive TCC After Treatment With an Immune Checkpoint Inhibitor
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding was withdrawn prior to first enrollment.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000022801
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Transitional Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — pembrolizumab; Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pembrolizumab and Ramucirumab (Experimental): Patients with progressive transitional cell carcinoma after treatment with an immune checkpoint inhibitor will receive Pembrolizumab and Ramucirumab.
  Interventions: Drug: Pembrolizumab and Ramucirumab

INTERVENTIONS:
Drug: Pembrolizumab and Ramucirumab — Patients will receive Pembrolizumab 200 mg & Ramucirumab 10 mg/kg every 3 weeks.

SUMMARY:
This study is designed to evaluate response and survival of treatment with the combination of pembrolizumab and ramucirumab in patients with progressive metastatic TCC after immune checkpoint inhibitor treatment.

DETAILED DESCRIPTION:
This is a phase II, non-randomized single center study designed to evaluate response and survival of treatment with the combination of pembrolizumab and ramucirumab in patients with progressive metastatic TCC after immune checkpoint inhibitor treatment.

The primary and secondary objectives are as follows:

Primary:

* Objective: To evaluate overall response rate (ORR) in patients treated with pembrolizumab and ramucirumab
* Hypothesis: The ORR will be ≥15% greater than the historical rate in published literature of patients treated with pembrolizumab alone

Secondary Objectives:

* Objective: To evaluate progression free survival (PFS) in patients treated with pembrolizumab and ramucirumab
* Hypothesis: The PFS will be ≥15% greater than the historical rate in published literature of patients treated with pembrolizumab alone
* Objective: To evaluate overall survival (OS) in patients treated with pembrolizumab and ramucirumab
* Hypothesis: The OS will be ≥15% greater than the historical rate in published literature of patients treated with pembrolizumab alone
* Objective: To evaluate differences in ORR, PFS and OS in patients treated with pembrolizumab and ramucirumab stratified by Bellmunt criteria.
* Hypothesis: Patients with high Bellmunt criteria scores will have lower rates of ORR, PFS and OS.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed transitional cell carcinoma of the urothelium (bladder, urethra, or renal pelvis). Patients with mixed pathology are eligible only if they have predominantly transitional cell tumor based on local pathology review.
2. Unresectable, locally advanced or metastatic disease.
3. Documented disease progression by RECIST 1.1 criteria to at least one prior line of systemic therapy and no more than three. Prior therapy for advanced disease must include an immune checkpoint inhibitor. Prior therapy in an adjuvant or neoadjuvant setting is not considered as a prior line of systemic chemotherapy, unless patient has rapidly progressed as defined by ≤ 6 months of last dose in this setting. If it is ≤ 6 months, it will be regarded as a prior line of treatment. Prior treatment with intravesicular chemotherapy, bacillus Calmette -Guérin (BCG), or platinum given as a radiation-sensitizing agent will not be considered as a systemic line of treatment.
4. A brain scan via CT with contrast or MRI is to be performed to confirm absence of intracranial metastasis.
5. The presence of measurable disease based on the Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1) as determined by the site study team. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.

   a. Measurable disease must still be present after pretreatment core-needle or excisional biopsy.
6. Provided signed informed consent and are amenable to compliance with protocol schedules and testing.
7. Provided tissue for biomarker analysis from a newly obtained core or excisional biopsy of a tumor lesion using a non-significant risk procedure prior to enrollment. Repeat samples may be required if adequate tissue is not provided.
8. ECOG Performance Status of 0 or 1.
9. Age: 18 years of age or older on day of signing consent.
10. Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures.
11. The patient's urinary protein is ≤1+ on dipstick or routine urinalysis (UA; if urine dipstick or routine analysis is ≥2+, a 24-hour urine collection for protein must demonstrate <1000 mg of protein in 24 hours to allow participation in this protocol)
12. Adequate organ function, as defined in the table below, with all screening labs performed within 14 days of treatment initiation:
13. Patients on full-dose anticoagulation must be on a stable dose (minimum duration 14 days) of oral anticoagulant or low molecular weight heparin. If receiving warfarin, the patient must have an INR ≤ 3.0 and no active bleeding (i.e., no bleeding within 14 days prior to first dose of study treatment) or pathological condition present that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices). Patients on anticoagulation therapy with unresected primary tumors or local tumor recurrence following resection are not eligible.
14. An anticipated life expectancy of ≥3 months.
15. Resolution, except where otherwise stated in the inclusion criteria, of all clinically significant toxic effects of prior systemic cancer therapy, surgery, or radiotherapy to Grade ≤1 by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0 (v 5.0)
16. For male patients, are sterile (including vasectomy confirmed by post-vasectomy semen analysis) or agree to use a reliable method of birth control and to not donate sperm during the study and for at least 120 days following the last dose of study treatment. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
17. For female patients, are surgically sterile, are postmenopausal, or agree to use a highly effective method of birth control (2 methods preferred) during the study and for 120 days following the last dose of study treatment.
18. If female and of childbearing potential, must have a negative serum or urine pregnancy test within 7 days prior to enrollment.

Note: Non-childbearing potential (by other than medical reasons). Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.

Exclusion Criteria:

1. Have non-measurable disease
2. Have known brain metastases, uncontrolled spinal cord compression, or leptomeningeal disease
3. Have received ≥3 lines of prior systemic anticancer therapy for advanced disease in urothelial cancer patients
4. Have a serious illness or medical condition(s) including, but not limited to, the following:

   1. Diagnosis of immunodeficiency or are receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. The use of physiologic doses of corticosteroids may be approved after evaluation by the Sponsor-Investigator.
   2. Active autoimmune disease that has required systemic treatment in past 2 years (that is, with use of disease-modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (for example, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
   3. Received a prior autologous or allogeneic organ or tissue transplantation
   4. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
   5. History of interstitial lung disease
   6. Known human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)-related illness
   7. Known active Hepatitis B or Hepatitis C infection
   8. Liver cirrhosis at a level of Child-Pugh B (or worse)
   9. Liver cirrhosis (any degree) and a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis. Clinically meaningful ascites is defined as ascites resulting from cirrhosis and requiring ongoing treatment with diuretics and/or paracentesis.
   10. Have a serious cardiac condition, such as congestive heart failure; unstable angina pectoris; myocardial infarction within the last 6 months; valvulopathy that is severe, moderate, or deemed clinically significant; or arrhythmias that are symptomatic or require treatment (not including patients with rate-controlled atrial fibrillation)
   11. Active or uncontrolled clinically serious infection
5. The patient is pregnant or breast-feeding.
6. The patient has radiologically documented evidence of major blood vessel invasion or encasement by cancer.
7. Known psychiatric or substance abuse disorders
8. Known allergy or hypersensitivity reaction to any of the treatment components
9. History of hematologic malignancy, malignant primary brain tumor, malignant sarcoma, or other malignant priory solid tumor not under study, except:

   1. no evidence of that disease for 5 years
   2. adequately treated non-melanoma skin cancer
   3. curatively treated cervical carcinoma in situ or other noninvasive carcinoma or in situ neoplasm
10. Have received any previous systemic therapy (including investigational agents) targeting VEGF/VEGF receptor. Prior therapy with anti-CD137 or anti-CTLA-4 antibody is permitted.
11. Have received a live vaccine within 30 days prior to enrollment Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
12. Have received transfusion of blood products (including platelets or red blood cells) or administration of colony-stimulating factors (including granulocyte colony-stimulating factor [G-CSF], granulocyte-macrophage colony-stimulating factor [GM-CSF], or recombinant erythropoietin) within 4 weeks prior to Cycle 1 Day 1
13. Have a significant bleeding disorder or vasculitis or had a Grade ≥3 bleeding episode within 12 weeks prior to enrollment
14. Have experienced any arterial thrombotic event, including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack, within 6 months prior to enrollment
15. Have experienced any Grade 3 or 4 venous thromboembolic event (VTE) that is considered by the investigator to be life threatening or that is symptomatic and not adequately treated by anticoagulation therapy, within 6 months prior to enrollment
16. Have a history of gastrointestinal perforation and/or fistula within 6 months prior to enrollment or risk factors for perforation.
17. Have a bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection (hemicolectomy or extensive small intestine resection, either condition with chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea
18. Have uncontrolled hypertension, as defined as Grade >2 CTCAE Version 5.0 (clinically, the patient continues to experience elevated blood pressure [systolic >160 mmHg and/or diastolic >100 mmHg] despite medications)
19. Are receiving chronic therapy with any of the following within 7 days prior to enrollment (note: aspirin use at doses up to 325 mg/day is permitted):

    1. nonsteroidal anti-inflammatory agents (NSAIDs; such as indomethacin, ibuprofen, naproxen, or similar agents)
    2. other anti-platelet agents (such as clopidogrel, ticlopidine, dipyridamole, or anagrelide)
20. Have had a serious or non-healing wound, ulcer, or bone fracture within 28 days prior to enrollment
21. Have an elective or a planned major surgery during the course of the trial or has undergone major surgery within 28 days prior to enrollment, or central venous access device placement within 7 days prior to enrollment. Note: If patient received major surgery, the patient must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
22. Have had chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks and/or monoclonal antibody treatment within 4 weeks prior to enrollment or not recovered (that is, ≤ Grade 1 or at baseline) from previously administered agents. Note: Neuropathy (≤ Grade 2) or nonserious and nonlife-threatening toxicities, such as alopecia, altered taste, or nail changes, are an exception to this criterion. Note: Palliative radiotherapy during the study, if clinically indicated, can be considered after consultation with the medical monitor.
23. Are currently enrolled in a clinical trial involving an investigational product or non-approved use of a drug, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study or discontinued study drug within 28 days or 5 half-lives of the drug, whichever is longer, prior to enrollment. Patients participating in surveys or observational studies are eligible to participate in this study.
24. Are or have an immediate family member (for example, spouse, parent/legal guardian, sibling, or child) who is investigational site or sponsor staff directly involved with this trial, unless prospective institutional review board (IRB) approval (by chair or designee) is given allowing exception to this criterion for a specific patient
25. Have radiographic evidence of intratumor cavitation
26. Have a history of gross hemoptysis (defined as bright red blood or ≥1/2 teaspoon) within 2 months prior to enrollment
27. Have pleural effusion, pericardial fluid, or ascites requiring drainage every other week or more frequently
28. Have superior vena cava syndrome
29. Have preexisting idiopathic pulmonary fibrosis as evidenced by CT scan/X-ray at baseline; have or had any disease of acute lung injury, idiopathic pulmonary fibrosis, or pneumoconiosis evident on an X-ray; have or had any disease of radiation pneumonia or drug-induced pneumonia.
30. Has a known history of active TB (Bacillus Tuberculosis).
31. Unable to have a pretreatment core-needle or excisional biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 24 months
  The objective overall response rate (ORR) is the proportion of enrolled patients who have received any amount of either study drug, have at least 1 post baseline tumor image, and achieve a best overall response of complete response (CR) or partial response (PR). The ORR will be assessed based on RECIST 1.1 and irRECIST.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to 24 months
  Progression-free survival (PFS) is defined as the time from the date of first study treatment until the date of the first observed radiographically documented PD or death due to any cause, whichever is earlier.
Overall survival (OS) | Up to 24 months
  Overall survival (OS), including 1- and 2- year survival rates, is determined from the date of first study treatment until death due to any cause. If the patient was alive at the data inclusion cutoff date for the analysis (or was lost to follow-up), OS will be censored on the last date the patient was known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hurwitz, PhD, MD, Principal Investigator — Assistant Professor of Medicine (Medical Oncology) Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No